CLINICAL TRIAL: NCT01346722
Title: Absorption of Zinc From Mixed Diets Containing Conventional Bangladeshi Rice, Zinc-biofortified Bangladeshi Rice, or Conventional Bangladeshi Rice With Added Zinc Among Young Children in a Peri-urban Community
Brief Title: Zinc Absorption From Zinc Biofortified Rice
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: HarvestPlus (Other); International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2008-046
Record Dates: First submitted 2011-04-27; First posted 2011-05-03 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2011-05

CONDITIONS: Malnourished Children
MeSH Terms: interventions — zinc(II) chromium(III) hydroxide 2,2'-azino-di-(3-ethylbenzothiazoline)-6-sulfonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): zinc biofortified rice-based diet (Diet-ZBfR) will be compared with conventional rice-based diet (Diet- CR)
  Interventions: Other: Diet-ZnBfR; Other: Diet- CR
- Group B (Other): zinc biofortified rice-based diet (Diet-ZBfR) will be compared with a rice-based diet plus zinc fortificant (Diet-CR+Z)
  Interventions: Other: Diet-ZnBfR; Other: CR + Zn

INTERVENTIONS:
Other: Diet-ZnBfR — zinc biofortified rice-based diet
  Arms: Group A
Other: Diet- CR — conventional rice-based diet
  Arms: Group A
Other: Diet-ZnBfR — zinc biofortified rice-based diet
  Arms: Group B
Other: CR + Zn — conventional rice-based diet plus zinc fortificant (Diet-CR+Z).
  Arms: Group B

SUMMARY:
a. To measure the amount of zinc absorbed from ZnBfR compared with the amount absorbed from CR and from CR fortified with added zinc, using the triple stable isotope tracer ratio technique in young children.

Methods:

Investigators will measure the amount of zinc absorbed from ZnBfR compared to that absorbed from a conventional Bangladeshi rice (Diet-CR) (control). They will also compare the zinc absorption from ZnBfR with that from zinc-fortified conventional rice (Diet-CR+Z). The study will be a cross-over, randomized, controlled clinical study. Forty-four children aged 36-59 mo of either sex will be recruited from the same community as mentioned before, and participants will be individually randomized, in equal numbers, to one of the two comparison groups, A and B. During an initial one-day acclimatization period, the participants will receive the conventional rice-based diet three times a day, to confirm that participants will accept the study diets and adhere to the study procedures. On study days 2 and 4, in comparison group A, participants will receive either the Diet-ZBfR or Diet-CR based on the random assignments, and participants will receive Diet-CR or Diet ZBfR, respectively, on days 3 and 5 (i.e., the diet not received on days 2 and 4), Likewise, in comparison group B, the participants will receive either Diet-ZBfR or Diet-CR+Z on days 2 and 4 based on the random assignments, and participants will receive Diet-CR+Z or the Diet-ZBfR, respectively, on days 3 and 5 (i.e., the diet not received on days 2 and 4). Investigators will use zinc stable isotope tracer techniques to measure the fractional absorption of zinc, in which tracer:tracee ratios will be measured in spot urine samples following administration of an intravenously administered tracer (68Zn) and one of two oral tracers (70Zn, 67Zn) provided with test meals over a four-day period.

Outcome measures/variables:

Intake of total dietary zinc (TDZ) and phytate for each subject will be calculated during the clinical study. Fractional absorption of zinc (FAZ) will be determined from the isotopic ratios obtained in urine samples using the following equation, which shows, as an example, the calculation that will be used for zinc absorption from the diet traced with 67Zn:

FAZ = 67Zn tracer:tracee ratio / 68Zn tracer:tracee ratio * (68Zn dose given IV / 67Zn dose given orally)

Total absorbed zinc (TAZ) for each child will be calculated as follows:

TAZ (mg/d) = TDZ (mg/d) * FAZ

DETAILED DESCRIPTION:
It is well documented that zinc supplementation to low-income population results in the reduced incidence of childhood diarrhoea and pneumonia, and improves growth of stunted children. In Bangladesh, the risk of zinc deficiency is considered to be high and children could benefit greatly by improving their zinc intakes on a daily basis. Zinc supplementation at a national scale would be a formidable task. There is a need to find an alternative. It might be sustainable to improve intake of zinc through fortified staples, e.g. rice with increased amounts of zinc; in fact such biofortified rice has been developed through conventional breeding, which is designed to contain an amount of zinc that could meet at least 40% of the daily requirement.

In the first round of the previously approved and completed studies, total absorbed zinc (TAZ) did not differ when diets containing zinc biofortified rice (ZnBfR) or conventional rice (CR) were compared. Thus, the investigators plan to repeat this study using a new variety of (ZnBfR)that is expected to have higher zinc content than the variety previously studied. Initially, the investigators will also conduct a pilot study in 4 subjects using a modified isotope administration protocol such that the oral tracers will be given on two days each at half the original dose each day so as to provide a lower proportion of the total daily zinc intake as tracer solution.

Hypotheses:

1. Young children will have greater total absorbed zinc (TAZ) when participants consume mixed diets containing ZnBfR than when participants consume the same diets containing CR.
2. TAZ will not differ in children who receive the ZnBfR-containing diet or the same diet containing CR plus sufficient additional zinc to match the zinc content of the ZnBfR diet.

Objectives:

1. To measure the amount of zinc absorbed from ZnBfR compared with the amount absorbed from CR and from CR fortified with added zinc, using the triple stable isotope tracer ratio technique in young children.
2. To assess the intestinal function of the children, using a sugar permeability test (lactulose:mannitol test).
3. (Pilot study) To verify that the modified tracer dose will provide adequate signal for assessing zinc absorption.

Methods:

To assess the potentials for biofortified rice in providing a good, bioavailable source of additional zinc, the investigators propose to measure zinc absorption from rice-based meals among Bangladeshi preschool children. The investigators will measure the amount of zinc absorbed from ZnBfR compared to that absorbed from a conventional Bangladeshi rice (Diet-CR) (control). The investigators will also compare the zinc absorption from biofortified rice with that from zinc-fortified conventional rice (Diet-CR+Z). The study will be a cross-over, randomized, controlled clinical study. Initially, a pilot study will be conducted with a modified dose of zinc stable isotope among 4 children aged 36-59 months of either sex from a peri-urban community in Dhaka. Later on, 44 children aged 36-59 months of either sex will be recruited from the same community as mentioned before, and participants will be individually randomized, in equal numbers, to one of the two comparison groups, A and B. During an initial one-day acclimatization period, the study children will receive the conventional rice based diet three times a day, to confirm that participants will accept the study diets and adhere to the study procedures. On study days 2 and 4, in comparison group A, the study subjects will receive either the Diet-ZBfR or Diet-CR based on the random assignments, and participants will receive Diet-CR or Diet ZBfR, respectively, on days 3 and 5 (i.e., the diet not received on days 2 and 4), Likewise, in comparison group B, the study subjects will receive either Diet-ZBfR or Diet-CR+Z on days 2 and 4 based on the random assignments, and participants will receive Diet-CR+Z or the Diet-ZBfR, respectively, on days 3 and 5 (i.e., the diet not received on days 2 and 4). The investigators will use zinc stable isotope tracer techniques to measure the fractional absorption of zinc, in which tracer : tracee ratios will be measured in spot urine samples following administration of an intravenously administered tracer (68Zn) and one of two oral tracers (70Zn, 67Zn) provided with test meals over a four-day period.

Outcome measures/variables:

Intake of total dietary zinc (TDZ) and phytate for each subject will be calculated during the clinical study. Fractional absorption of zinc (FAZ) will be determined from the isotopic ratios obtained in urine samples using the following equation, which shows, as an example, the calculation that will be used for zinc absorption from the diet traced with 67Zn:

FAZ = 67Zn tracer:tracee ratio / 68Zn tracer:tracee ratio * (68Zn dose given IV / 67Zn dose given orally)

Total absorbed zinc (TAZ) for each child will be calculated as follows:

TAZ (mg/d) = TDZ (mg/d) * FAZ

ELIGIBILITY:
Inclusion Criteria:

* Age: 42 children aged 36-59 mo; Either sex
* WLZ and HAZ: >-2 Z-Score
* No longer breastfed
* No H/O diarrhoea in last 14 days
* Given anti-helminthics in last three months

Exclusion Criteria:

* Not meeting the inclusion criteria

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Total absorbed zinc | 10 days
  Total absorbed zinc (TAZ) for each child will be calculated as follows:
  TAZ (mg/d) = Total Dietray Zinc (TDZ) (mg/d) * Frcational Absorbed Zinc (FAZ)

CONTACTS AND LOCATIONS:
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Islam MM, Woodhouse LR, Hossain MB, Ahmed T, Huda MN, Ahmed T, Peerson JM, Hotz C, Brown KH. Total zinc absorption from a diet containing either conventional rice or higher-zinc rice does not differ among Bangladeshi preschool children. J Nutr. 2013 Apr;143(4):519-25. doi: 10.3945/jn.112.169169. Epub 2013 Feb 20. PMID 23427330